CLINICAL TRIAL: NCT07197710
Title: Assessing the Efficacy of Imagined Acupuncture for Postoperative Acute Pain Management in Spinal Surgery
Brief Title: Imagined Acupuncture for Postoperative Pain After Spinal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jingping Wang, MD, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Jingping Wang, MD, Ph.D., Associate Professor Staff Anesthesiologist & Pain Physician, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025P001674
Record Dates: First submitted 2025-09-25; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pain Management
Keywords: Postoperative Acute Pain; Imagined Acupuncture
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Imagined Acupuncture Intervention (Experimental): Participants assigned to Group 1 will receive standard postoperative care and a daily VGAIT session once per day for seven consecutive days following surgery. Each session will last approximately 30 minutes and will be guided by a standardized video designed to induce acupuncture imagery and mental engagement. VGAIT will be administered at the same time each day (e.g., 9:00 AM ± 30 minutes). VAS and ODI assessments will be administered following the completion of the video session. The initial video session will be administered once the patient has fully regained consciousness in the post-anesthesia care unit (PACU) following surgery.
  Interventions: Other: video-guided acupuncture imagery treatment (VGAIT)
- Group 2: Education video (Sham Comparator): Participants in the control group will receive standard postoperative care and Education video without any simulated acupuncture intervention. VAS and ODI assessments will be conducted at the same intervals as in Group 1 for consistency and comparison.
  Interventions: Other: Education video

INTERVENTIONS:
Other: video-guided acupuncture imagery treatment (VGAIT) — Unlike traditional acupuncture, VGAIT can be self-administered and does not require physical needle insertion, making it a practical alternative for patients seeking non-invasive pain management.
  Arms: Group 1: Imagined Acupuncture Intervention
Other: Education video — Education video about postoperative precautions
  Arms: Group 2: Education video

SUMMARY:
The goal of this clinical trial is to evaluate whether imagined acupuncture can reduce postoperative acute pain in adult patients undergoing spinal surgery. The main questions it aims to answer are:

Does video-guided imagined acupuncture improve postoperative pain control?

Does the intervention reduce opioid consumption and improve functional recovery in the immediate postoperative period?

Researchers will compare the imagined acupuncture group to the control education video group to see if imagery-based intervention leads to better pain outcomes and reduced analgesic use.

Participants will:

Watch a 30-minute video once daily for 7 consecutive days after surgery

Complete pain and function assessments during the hospital stay and postoperative follow-up

ELIGIBILITY:
Inclusion Criteria:

* Undergoing 1- to 2-level primary spine surgery
* Aged 18 years or older
* Willing and able to receive postoperative imagined acupuncture (VGAIT)
* Able to provide written informed consent

Exclusion Criteria:

* Undergoing revision surgery or procedures involving more than 3 spinal levels
* History of prior spinal surgery
* Intraoperative complications likely to interfere with postoperative pain assessment
* Diagnosed with severe cognitive impairment or psychiatric disorders that impair participation or communication
* Pregnant or breastfeeding
* Unable to cooperate with treatment or pain assessments Individuals with uncorrectable vision impairment that would interfere with viewing study videos or completing study questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-19 (Estimated); Study Completion 2026-09-19 (Estimated)

PRIMARY OUTCOMES:
Pain Scores (VAS) | During the first postoperative week (Days 0-6)
  Pain intensity will be assessed using the Visual Analog Scale (VAS) daily, including VAS at rest, VAS on movement
2) Functional Scores (ODI) | On postoperative Day6
  Functional status will be evaluated using the Oswestry Disability Index (ODI)
3) Rescue Opioid Consumption | On postoperative Day6
  The total amount of rescue opioid medication used during the first postoperative week will be recorded in milligrams (oral and intravenous)

SECONDARY OUTCOMES:
1) Time to First Rescue Analgesia | On postoperative Day6
  The exact time (in hours and minutes) from the end of surgery to the administration of the first rescue analgesic will be recorded
2) Total Analgesic Consumption | On postoperative Day6
  The cumulative amount of all pain medications (opioid and non-opioid, oral and intravenous) administered within 7 days postoperatively, recorded in milligrams.
3) Length of Hospital Stay | On postoperative Day6
  Measured as the number of days from the date of surgery to the date of hospital discharge.
4) Adverse Effects | On postoperative Day6
  Incidence of treatment-related side effects, including nausea, vomiting, dizziness, respiratory depression, urinary retention, ileus, or any other reported complications.
5) Additional Assessment Tools | On postoperative Day6
  RCSQ: Richards-Campbell Sleep Questionnaire

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns about patient privacy and the sensitive nature of the data collected, including postoperative pain scores and behavioral intervention responses.

REFERENCES:
- [Background] Kong J, Eshel MN. Applying the Power of the Mind in Acupuncture Treatment of Pain. Med Acupunct. 2020 Dec 1;32(6):367-372. doi: 10.1089/acu.2020.1477. Epub 2020 Dec 16. PMID 33362889
- [Background] Kong J, Kaptchuk TJ, Polich G, Kirsch I, Vangel M, Zyloney C, Rosen B, Gollub RL. An fMRI study on the interaction and dissociation between expectation of pain relief and acupuncture treatment. Neuroimage. 2009 Sep;47(3):1066-76. doi: 10.1016/j.neuroimage.2009.05.087. Epub 2009 Jun 6. PMID 19501656
- [Background] Cao J, Tu Y, Orr SP, Wilson G, Kong J. Modulatory Effects of Actual and Imagined Acupuncture on the Functional Connectivity of the Periaqueductal Gray and Ventral Tegmental Area. Psychosom Med. 2021 Oct 1;83(8):870-879. doi: 10.1097/PSY.0000000000000984. PMID 34292206
- [Background] Cao J, Tu Y, Orr SP, Lang C, Park J, Vangel M, Chen L, Gollub R, Kong J. Analgesic Effects Evoked by Real and Imagined Acupuncture: A Neuroimaging Study. Cereb Cortex. 2019 Jul 22;29(8):3220-3231. doi: 10.1093/cercor/bhy190. PMID 30137262
- [Background] Cao J, Tu Y, Wilson G, Orr SP, Kong J. Characterizing the analgesic effects of real and imagined acupuncture using functional and structure MRI. Neuroimage. 2020 Nov 1;221:117176. doi: 10.1016/j.neuroimage.2020.117176. Epub 2020 Jul 17. PMID 32682992
- [Background] Kong Q, Sacca V, Walker K, Hodges S, Kong J. Thalamocortical Mechanisms Underlying Real and Imagined Acupuncture. Biomedicines. 2023 Jun 26;11(7):1830. doi: 10.3390/biomedicines11071830. PMID 37509469
- [Background] Cao J, Orr SP, Wilson G, Kong J. Imagined and Actual Acupuncture Effects on Chronic Low Back Pain: A Preliminary Study. Neural Plast. 2020 Jul 1;2020:8579743. doi: 10.1155/2020/8579743. eCollection 2020. PMID 32684925